CLINICAL TRIAL: NCT02971163
Title: SynDA: Syncope Decision Aid for Emergency Care
Brief Title: Syncope Decision Aid for Emergency Care
Acronym: SynDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GCO 15-1016; 1K23HL132052-01 (NIH)
Record Dates: First submitted 2016-11-16; First posted 2016-11-22 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Syncope
Keywords: Syncope; Shared Decision-Making; Emergency Medicine; Decision Aid
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SynDA (Experimental): The research coordinator will print the appropriate version of the SynDA based on the patient's individualized risk score and the corresponding estimated probability of a serious medical event within 30 days.
  Interventions: Behavioral: SynDA
- Control (No Intervention): Patients in the control arm will receive usual emergency care pertaining to syncope.

INTERVENTIONS:
Behavioral: SynDA — SynDA is a paper-based, personalized decision aid which gives information to patients about their medical condition (i.e. syncope), future risk, and options for care. It is written in lay language and aims to create an informed conversation between a patient and their ED provider.
  Other Names: Syncope Decision Aid
  Arms: SynDA

SUMMARY:
Syncope, or transient loss of consciousness/fainting, is a common emergency department (ED) complaint responsible for over 1 million ED visits yearly. Potential causes include benign conditions such as dehydration or vaso-vagal syncope. Rarely, syncope is the result of serious cardiac conditions. In older patients without a clear cause of syncope hospital admission is frequently initiated at very low risk thresholds, though there is little evidence that these admissions improve patient outcomes. These decisions are often made without significant patient input or discussion of reasonable alternatives. In this situation, a patient's values, preferences, and particular circumstances should be taken into account. This mutualistic approach to clinical management is referred to as Shared Decision-Making. Shared Decision-Making (SDM) is a joint process of choice selection between providers and patients in clinical scenarios where multiple reasonable management options exist. To improve syncope emergency care, the researchers can leverage recent advances in risk stratification to engage patients in SDM and deliver superior, patient-centered care.

This study will provide the groundwork for a larger, randomized controlled trial evaluating the effects of the decision aid for management of low-risk syncope.

DETAILED DESCRIPTION:
Setting:

Mount Sinai Hospital (MSH) has a 61-bed adult Emergency Department with a volume of over 100,000 patient visits/year or approximately 300 visits/day. MSH is a large academic tertiary care medical center located in East Harlem and serves a large black and Hispanic community.

Projected Recruitment: There are approximately 60 MSH ED visits for syncope per month of which 35 per month are by patients above age 30. Roughly half of these do not have a clear etiology of their syncope discovered in the ED. The researchers project that of the 17 potentially eligible patients per month, three will be successfully enrolled for a projected 72 patient enrollees at the completion of the 24-month recruitment period. The PI, clinical research coordinators, and SRAs will monitor the real-time electronic tracking system for all ED patients and will identify any patient over age 30 with a chief complaint of syncope or loss of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department patient
* Age 30 years or above
* Chief complaint of syncope
* Capacity to make medical decisions
* Speak and read English
* Working phone number and fixed address

Exclusion Criteria:

* Altered Mental Status
* Cognitive Impairment
* Serious acute diagnosis:

  (e.g. clinically significant cardiac dysrhythmia, structural heart disease, gastrointestinal hemorrhage, myocardial infarction, pulmonary embolism, pneumonia, arterial dissection, serious infection, ectopic pregnancy, subarachnoid hemorrhage, or stroke.)
* Hemodynamic instability
* Inability to read or speak English
* Major communication barrier
* Lack of phone number or fixed address
* Too high risk as per physician judgment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01; Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Richardson, MD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Probst MA, Lin MP, Sze JJ, Hess EP, Breslin M, Frosch DL, Sun BC, Langan MN, Thiruganasambandamoorthy V, Richardson LD. Shared Decision Making for Syncope in the Emergency Department: A Randomized Controlled Feasibility Trial. Acad Emerg Med. 2020 Sep;27(9):853-865. doi: 10.1111/acem.13955. Epub 2020 Apr 2. PMID 32147870

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After screening 351 patients, 51 randomized, one was excluded because not syncope, resulting in 50 participants enrolled with unexplained syncope from January 2017 to January 2019.
Period: Overall Study
Arm/Group | SynDA | Control
Started | 24 | 26
Completed | 20 | 24
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SynDA | Control | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54.5 [45.3 to 70] | 60 [47.8 to 73] | 58.5 [46.3 to 71.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 12 | 9 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African-American | 7 | 11 | 18
  Hispanic/Latino | 5 | 5 | 10
  White | 10 | 7 | 17
  Asian | 0 | 1 | 1
  Other | 2 | 2 | 4
Control Preferences Scale [Count of Participants; unit: Participants] — A validated single question measure of patient's desire for involvement in medical decisions that ranges from 1 (active) to 3 (collaborative) to 5 (passive).
  Participants
    1 | 3 | 0 | 3
    2 | 8 | 7 | 15
    3 | 10 | 13 | 23
    4 | 2 | 2 | 4
    5 | 0 | 2 | 2
    Missing data | 1 | 2 | 3
Subjective Numeracy Score (SNS) [Mean (Standard Deviation); unit: units on a scale] — The SNS consists of three questions summed to give a min and max score of 3-18 with higher scores indicating higher subjective numeracy skills.
  units on a scale | 13.2 (2.6) | 12.6 (2.6) | 12.9 (2.6)
Short Literacy Survey (SLS) [Mean (Standard Deviation); unit: units on a scale] — The SLS consists of three questions summed to give a score of 3-15 with higher scores indicating greater subjective health literacy.
  units on a scale | 13.2 (2.6) | 12.6 (2.6) | 12.9 (2.6)
Education [Count of Participants; unit: Participants]
  Some High School | 1 | 1 | 2
  High School Graduate/GED | 3 | 4 | 7
  Some College | 8 | 7 | 15
  College Graduate | 4 | 6 | 10
  Graduate School | 8 | 8 | 16
Income [Count of Participants; unit: Participants]
  Less than $20,000 | 2 | 7 | 9
  $20,000 to $29,999 | 1 | 4 | 5
  $30,000 to $39,999 | 2 | 2 | 4
  $40,000 to $59,999 | 3 | 2 | 5
  $60,000 to $79,999 | 3 | 0 | 3
  $80,000 to $99,999 | 2 | 1 | 3
  $100,000 or more | 4 | 5 | 9
  Rather Not Say | 7 | 5 | 12
Canadian Syncope Risk Score [Count of Participants; unit: Participants]
  Low: 0 (≈2% risk) | 3 | 6 | 9
  Medium: 1 (≈3% risk) | 13 | 15 | 28
  Medium: 2 (≈5% risk) | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants at End of Study
Description: Feasibility of the study will be measured by the number of participants successfully enrolled at the end of the study period.
Time Frame: Two years
Measure: Count of Participants; unit: Participants
Arm/Group | SynDA | Control
Number analyzed (Participants) | 24 | 26
Participants | 20 | 24

2. Secondary Outcome: Patient Knowledge
Description: One brief post-encounter survey will be given to the patient to assess their knowledge surrounding syncope and their satisfaction with their care during the ED visit. Scores full range is 0-9, higher score indicates more knowledge
Time Frame: Within 2 hours post ED disposition on Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SynDA | Control
Number analyzed (Participants) | 24 | 26
score on a scale | 5.2 (1.8) | 5.3 (1.8)

3. Secondary Outcome: Decisional Conflict Scale
Description: Decisional quality will be measured by administering the Decisional Conflict Scale to all patients after disposition decision has been made. The decisional conflict scale total score range from 0 (no decisional conflict) to 10 (extremely high decisional conflict).
Time Frame: Within 2 hours post ED disposition on Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SynDA | Control
Number analyzed (Participants) | 24 | 26
score on a scale | 8.9 (1.5) | 9 (1.6)

4. Secondary Outcome: Utilization Outcomes
Description: Number of patients admitted to the hospital or sent to observation unit at index visit and number of patients admitted to the hospital, or had an office visit or during 30-day follow-up period
Time Frame: Day 1 and 30 day follow up period
Measure: Count of Participants; unit: Participants
Arm/Group | SynDA | Control
Number analyzed (Participants) | 24 | 26
Participants
  Admitted to hospital Day 1 | 0 | 0
  Sent to observation unit Day 1 | 4 | 7
  Admitted to hospital 30 day follow up period | 1 | 1
  Office visit 30 day follow up period | 14 | 17

5. Secondary Outcome: Number of Participants With Repeat Visits to the ED
Description: Number of participants with repeat visits to the ED during 30-day follow-up period
Time Frame: 30-day follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | SynDA | Control
Number analyzed (Participants) | 20 | 24
Participants | 1 | 2

6. Secondary Outcome: Participants With New Significant Clinical Diagnosis
Description: Number of participants with clinical diagnosis at 30 days after index visit to the ED
Time Frame: at 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SynDA | Control
Number analyzed (Participants) | 20 | 24
Participants
  Acute Stroke | 1 | 0
  Heart Failure | 1 | 0
  Cardiac Arrhythmia | 0 | 1
  Large Pericardial Effusion | 0 | 1

7. Secondary Outcome: Number of Diagnostic Testing
Description: Number of diagnostic test (which may include but not limited to exercise stress testing, echocardiography, computed tomography scans) performed
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | SynDA | Control
Number analyzed (Participants) | 24 | 26
Participants | 1 | 1

8. Secondary Outcome: OPTION-5 Scale
Description: The degree of patient involvement in the disposition decision as measured by the OPTION (observing patient involvement in decision making) scale. The OPTION-5 scale is a brief, 5-item instrument used by a trained observer to measure the degree of patient involvement in clinical decision-making and has demonstrated validity and reliability. Full scores range from 0 to 100, with higher scores indicating higher levels of patient involvement.
Time Frame: up to 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SynDA | Control
Number analyzed (Participants) | 24 | 26
score on a scale | 52.0 (18) | 26.6 (21)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | SynDA | Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

LIMITATIONS AND CAVEATS:
Small sample size of only English-speaking patients from a single, busy, urban, academic center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02971163/Prot_SAP_000.pdf